CLINICAL TRIAL: NCT06491277
Title: The Effect of Ankle Floss Band Application on Balance, Proprioception and Performance
Brief Title: The Effect of Ankle Floss Band on Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, PHD, Physiotherapist,Thesis Advisor, Alanya Alaaddin Keykubat University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023/01
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Ankle Instability
Keywords: physical Functional performance; Floosband; Bandage
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flossband Group (Active Comparator): Our study began by applying flossband to the football players. The players were first assessed without the flossband, and then reassessed with the flossband to measure its effectiveness. This group was referred to as the 'Study Group.'
  Interventions: Other: Flossband
- Controlled Group (Sham Comparator): After the specified rest period, the football players were evaluated prior to the foam roller application. Seventy-two hours later, they were reassessed with the foam roller to measure the effectiveness of the application. This group was referred to as the 'Control Group.
  Interventions: Other: Controlled Group

INTERVENTIONS:
Other: Flossband — The use of Flossband (Sanctband COMPRE Floss 5.1 cm × 3.5 m; Sanct Japan Co., Ltd.), made of natural rubber, was applied starting from 5 cm below the ankle joint line with a 50% stretch. The band tension was increased to 70-75% around 2 cm above the attachment point of the Achilles tendon.
  Arms: Flossband Group
Other: Controlled Group — Cramer Tape Underwrap (7cm X 27m) foam bandage was applied starting 5 cm below the ankle joint line without tension. The control group received the same exercise protocol as the study group.
  Other Names: Sham
  Arms: Controlled Group

SUMMARY:
There is no study in the literature investigating the effects of ankle stimulation with the flossband soft tissue technique on balance and proprioception. The impact of flossband use on flexibility and static and dynamic balance in the lower extremities requires further research. It is likely that flossband, which has been found to enhance sports performance, also affects balance, proprioception, and performance. More research is needed to evaluate the benefits of flossband use on body movements and motor control. Therefore, the aim of this study is to evaluate the effects of flossband on balance, proprioception, and performance, given its known impact on sports performance.

DETAILED DESCRIPTION:
Objective: The aim of the study is to investigate the effects of exercises with flossband on balance, proprioception, and physical performance in the ankle.

Materials and Methods: Thirty-six football players were included in the study. As this was a serial group design the same football players were included in both the study group and the control group. There was a 72-hour break between the interventions for the study group and the control group. The study began with the study group. The study group received Flossband application while the control group received foam roller bandage application. The same exercises were conducted alongside both interventions. Measurements were taken before and after the interventions and exercises. Ankle dorsiflexion range of motion was evaluated using the weight-bearing lunge test, static balance using a smartphone application, dynamic balance using the Y-balance test, and proprioception using the joint position sense test. Additionally, the hop test was used to assess jumping performance.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25 years old.
* Engaged in regular football training for at least 3 years.

Exclusion Criteria:

* History of fractures and surgeries in the lower extremities.
* Diagnosed with other ankle and lower extremity problems.
* Presence of pain in the ankle and lower extremities.
* Systemic conditions such as deep vein thrombosis and embolism.
* Experience of pain during any measurement.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Football Players who plays in the man football team.
Enrollment: 36 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Weight Bearing Lunge Test | 3 days
  The ankle dorsiflexion range of motion was evaluated. Three tests were conducted for each participant, and the best score was recorded. Each assessment was performed before and after taping.
Static Balance Assesment | 3 days
  using the 'Accelerometer' application developed with Apple iPhone 14 and Dream Arc App Inventor, the static balance of football players was measured. Participants were instructed to stand on one leg for 30 seconds. Three trials were conducted, and the best score was recorded. The application recorded acceleration data in three axes (x, y, z) at a sampling rate of 20 Hz during the 30-second duration. Higher acceleration values indicated poorer balance.
Dynamic Balance Test | 3 days
  The Y balance test is a dynamic assessment widely used among athletes, requiring strength, flexibility, and proprioception, with good reliability. For the test, three equal-length strips of tape are placed on the floor to form a Y shape with angles of 90°, 135°, and 135° between them. The foot to be tested is placed at the intersection of the tapes, and the athlete is instructed to reach as far as possible in three different directions (anterior, posterolateral, posteromedial) while maintaining balance with the other foot. Football players attempted to reach maximum distance in each of these three directions, and these distances were recorded. The highest score from three successful reaches in each direction was normalized relative to leg length.Each assessment was performed before and after taping.
Proprioseptive Evaluation | 3 days.
  When evaluating joint position sense, the football player was seated on a chair with their feet flat on the ground and eyes closed. Using a smartphone goniometer application, the range of motion of both ankles was measured. The tested ankle was passively moved into a dorsiflexion position of 10 degrees and then returned to its original position. The player was asked to actively replicate the same position with their foot, and the deviation from the target 10 degrees was recorded. This process was repeated three times, and the average deviation was calculated.Each assessment was performed before and after taping
Triple Hop Test | 3 days
  This is a commonly used test for evaluating the functional abilities of the ankle and knee joints. The test measures the participant's balance, performance, and joint stability. A 6-meter scale is prepared, and the football player is instructed to stand on the assessed foot with arms by the sides and knees bent at a 45-degree angle in the starting position. The player is asked to perform three maximal forward jumps and land on the same line with the foot used for jumping. The distance between the heel and the starting point is measured, and the longest of two attempts is recorded.Each assessment was performed before and after taping

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat Üniversity, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No